CLINICAL TRIAL: NCT06679257
Title: Liquid Biopsies for Lung Allograft Damage Classification
Brief Title: Liquid biopsiEs fOr luNg AllogRaft Damage classificatiOn - LEONARDO
Acronym: LEONARDO
Status: Recruiting | Type: Observational
Sponsor: Jesper Magnusson (Other Government)
Responsible Party: Sponsor-Investigator, Jesper Magnusson, MD, PhD, Associate professor, Vastra Gotaland Region
Organization: Vastra Gotaland Region (Other Government)
Other Study IDs: LEONARDO
Record Dates: First submitted 2024-10-28; First posted 2024-11-07 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Lung Transplant Failure and Rejection; Lung Transplant Infection
MeSH Terms: conditions — Rejection, Psychology | interventions — Noninvasive Prenatal Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cell free DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lung transplanted patients: All eligible patients were transplanted and followed up within the catchment area of the participating centre.
  Interventions: Diagnostic Test: cell-free dNA

INTERVENTIONS:
Diagnostic Test: cell-free dNA — Blood samples taker per protocol, analyses performed by a lab blinded to the status of the respective patients

SUMMARY:
LTx has the shortest survival of all solid organ transplants. The complex and time-demanding diagnostics of allograft dysfunction are a significant reason for this.

The current study aims overarchingly to improve survival after lung transplantation (LTx) through precise and fast diagnostics. The specific aim is to develop direct-to-clinical implementation biomarkers for the most important aspects of long-term survival after LTx. An in-house-developed PCR-based cell-free-DNA methodology (cf-DNA) will be used for allograft damage and combined with specific other biomarkers to identify damage type. The current clinical golden standard for damage identification will be performed at every sampling instance.

The research will be a single-centre prospective observational cohort study. The control samples at all time points will consist of the samples without allograft damage. Blood will be drawn at fixed time points and clinical events. All analyses will be performed at a separate lab, blinded to the patient's status.

.

ELIGIBILITY:
Inclusion Criteria:

* Luing Transplanted and followed up within the reach of the study paricipating centres.

A good understanding to read and write within the languages in which the consent is provided.

Exclusion Criteria:

* Not Lung Transplanted or not followed up within the reach of the study paricipating centres.

No good understanding to read and write within the languages in which the consent is provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly lung transplanted patients within scandinavia
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Damage distinction | One month, three months, one year, three years, five years
  Null hypothesis: Levels of Cf-DNA is not different at samples taken with allograft damage and no allograft damage.

SECONDARY OUTCOMES:
Damage detection Limit | One month, three months, one year, three years, five years
  If the null hypothesis is disproven, measure optimal cut off for distincition beteween samples indicating damage and not indicating damage. Also distinction between different types of damage, finally if distinction is attainable trhough association wit other known biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes